CLINICAL TRIAL: NCT02356237
Title: The Effect of Episiotomy on Advanced Perineal Tears and Other Maternal and Fetal Outcomes - Randomized Controlled Multicentric Trial (EPITRIAL)
Brief Title: The Effect of Episiotomy on Maternal and Fetal Outcomes (EPITRIAL)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than expected recruitment rate, and larger than expected required sample.
Sponsor: Lena Sagi-Dain (Other)
Collaborators: Bnai Zion Medical Center (Other Government); Rambam Health Care Campus (Other); Hillel Yaffe Medical Center (Other Government); Ziv Medical Center (Other); The Baruch Padeh Medical Center, Poriya (Other Government); Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor-Investigator, Lena Sagi-Dain, Senior Obstetrician, Department of Obstetrics and Gynecology, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 125-14BNZ
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Anal Sphincter Injury
Keywords: Episiotomy; Obstetric Anal Sphincter Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No episiotomy (Experimental): Episiotomy will not be performed in this group. Deviation from protocol (i.e. episiotomy performance) will be allowed only according to the discretion of obstetrician in charge of the delivery, in cases of unequivocal benefit to the fetus.
  Interventions: Other: No episiotomy
- Selective episiotomy (No Intervention): The decision to perform episiotomy in this group will be based on routine delivery care, i.e. indistinguishable from any other delivery not participating in the trial.

INTERVENTIONS:
Other: No episiotomy — Avoidance of episiotomy
  Arms: No episiotomy

SUMMARY:
This study is aimed to evaluate the influence of episiotomy on various maternal and neonatal outcomes. Half of the participants will undergo selective episiotomy (according to routine delivery management at the particular hospital), while the other half will not undergo epitiotomy at all.

Our hypothesis is that no differences in maternal and neonatal outcomes will be demonstrated between these two groups.

DETAILED DESCRIPTION:
Episiotomy is one of the most prevalent surgical interventions at the delivery room, ranging in frequency from about 10% and up to 75%. The presumed benefits of this procedure include prevention of advanced (3rd and 4th degree) perineal tears, facilitation of fetal distress, easier suturing compared to that of spontaneous perineal tears, decreased postpartum pelvic organ injury including reduced risk of urinary and anal incontinence, and facilitation of labor in cases of shoulder dystocia. However, the cumulative evidence in the recent decades strongly points to the lack of episiotomy efficiency. Moreover, many studies indicate that episiotomy may be associated with increased maternal morbidity in terms of postpartum bleeding and pain, urinary incontinence and severe perineal tears. Cochrane Collaboration meta-analysis of randomized controlled trials has shown that selective episiotomy significantly decreases the risk of advanced perineal tears (relative risk of 0.67) and the overall need for perineal suturing (relative risk of 0.71), compared to routine episiotomy use. In addition, there is no uniform definition for the indications for episiotomy performance.

In accordance with literature evidence, we hypothesized that avoidance of episiotomy is not associated with increased risk of maternal and neonatal complications, compared to selective episiotomy use. Thus, the objective of our study is to compare maternal and neonatal outcomes in the group with no episiotomy performed to selective episiotomy use.

This randomized controlled clinical trial will be conducted in seven Northern public Israeli Hospitals from February 2015 to February 2019.

The following study protocol was constructed using consultation with experienced epidemiologist and several senior obstetricians.

Women fitting the inclusion criteria will receive a detailed explanation about the trial from one of the approved investigators and will carefully read the relevant forms. In case of agreement for participation in the study, informed consent form will be signed.

Each participant will undergo randomization into two groups:

1. Control group - in which the decision to perform episiotomy will be based on routine delivery care.
2. Study group - in which no episiotomy will be performed. Deviation from protocol and episiotomy performance in this group will be allowed only at the discretion of the obstetrician in charge of the delivery, only in cases of unequivocal benefit to the fetus.

The randomization will be carried out using computer software creating random numbers. Allocation to one of the two groups will be done at second stage of labor by opening of sealed opaque envelopes.

Mediolateral or lateral episiotomy (according to the accepted management in each medical center) will be performed during the crowning stage. The incision will be cut at an angle of 45-60º, for 3-4 cm of length.

Epidural anesthesia during labor will be administered in accordance with patient's request. Artificial rupture of membranes, augmentation of the contractions by oxytocin, the decision to perform vacuum extraction or a cesarean birth will be done at the discretion of the attending accoucher, in accordance with the accepted delivery management.

The following data will be obtained for each participant:

* Demographic and obstetric characteristics, including maternal age, weight, height and race, gestational age and pregnancy complications, clinical and sonographic estimated fetal weight.
* Delivery and neonatal parameters, including oxytocin use for labor augmentation and epidural anesthesia administration.
* Primary and secondary outcome measures (described elsewhere).

Sample size calculation was performed by a certified statistician with an extensive experience in clinical trials. It was based on the assumption that the worldwide rate of advanced perineal tears in the control group is 1.6% (according to the latest data reported at the annual Israeli Maternal and Fetal Medicine society meeting at November 2014), and that the rates of these tears in the study group is 1.072% (based on the above mentioned report of Cochrane Collaboration analysis, demonstrating relative risk of 0.67 with selective vs. routine episiotomy use). Given the confidence level of 95% and power of 80%, the required sample size is 14,842 (i.e. 7,421 women in each group).

A year after the trial initiation an interim analysis will be carried out, calculating the up-to-date rate of advanced perineal tears. Sample size will be recalculated based on this rate. In case of statistically significant difference in the primary outcome measure (advanced perineal tears) with a confidence level of 0.003, discontinuation of the trial will be considered due to demonstrated efficacy. Otherwise, the trial will be continued, and the required confidence level at the final statistical calculations will be 0.049.

At the end of data acquisition, statistical analysis will be carried out. Primary and secondary outcome measures will be compared between the two groups. In addition, the association between episiotomy characteristics (incision angle, length and distance from the initiation point to midperineum) to other outcome measures will be assessed.

Statistical analysis will be performed using SPSS software (SPSS Inc., Chicago, IL), in accordance with "intention to treat" concept. Data will be presented to the statistician in a blinded way, as groups "1" and "2", with non-disclosure of the number interpretation. Continuous variables will be presented as mean ± SD and compared using Student's t-test or Mann-Whitney test, as appropriate. Categorical data will be expressed as numbers (percentages) and compared using the Chi square test or Fisher's exact test, when appropriate. Relative risks with 95% confidence intervals will be calculated. A two tailed p<0.05 will be considered statistically significant for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Women in labor, or women scheduled for induction of labor, or women attending for a routine follow-up examination during third trimester of pregnancy.
* First vaginal delivery
* Singleton pregnancy above 34 gestational weeks
* Vertex presentation
* Women who are able to understand and sign the informed consent forms.

Exclusion Criteria:

Absolute contraindications for vaginal delivery (e.g. placenta previa, fetal macrosomia above 4.5 kg, genital herpes)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 676 (Actual)
Dates: Start 2015-06; Primary Completion 2018-05-06 (Actual); Study Completion 2018-05-06 (Actual)

PRIMARY OUTCOMES:
Obstetric Anal Sphincter injury | From the delivery to one hour after delivery
  Advanced (3rd and 4th degree) perineal tears, i.e. perineal lacerations involving the anal sphincter, diagnosed by a senior obstetrician

SECONDARY OUTCOMES:
1st and 2nd degree perineal tears | From the delivery to one hour after delivery
  1st and 2nd degree perineal tears i.e. lacerations not involving the anal sphincter), diagnosed by an attending accoucher immediately after delivery. Of note, episiotomy will be considered as a 2nd degree tear.
Duration of the second stage of labor | From beginning of full dilatation to the delivery of the baby
  Time in minutes from full dilatation stage of labor until the delivery of the baby
Postpartum hemorrhage | From delivery to one hour postpartum
  Excessive vaginal bleeding (above 500 ml according to the subjective evaluation of the attending accoucher, or associated with hemodynamic instability), from the moment of the delivery to one hour after delivery
Neonatal Apgar score | From the delivery to five minutes after delivery
  One and five minutes Apgar scores
Cord blood pH | From the delivery to first two minutes after delivery
  Cord blood pH - if measured
Need of any neonatal resuscitation procedures | From the delivery to one hour after delivery
  Any neonatal resuscitation procedures
Admission to Neonatal Intensive Care Unit (NICU) | From the delivery to one hour after delivery
  Admission to Neonatal Intensive Care Unit (NICU)
Shoulder dystocia | From the delivery of the head to the delivery of the shoulders or longer than 60 seconds interval between the delivery of the head to the delivery of the shoulders
  The occurrence of shoulder dystocia, defined as a requirement of obstetrical maneuvers for shoulder delivery, or longer than 60 seconds interval between the delivery of the head to the delivery of the shoulders
Episiotomy performance parameters (Indication for episiotomy performance) | During suturing (from the delivery to one hour after the delivery)
  Indication for episiotomy performance, incision characteristics - i.e. post-suture angle, length and initiation point of the incision, suturing accoucheur profession (midwife/obstetrician) and duration of his/her obstetric experience.
Characteristics of suturing procedure (The duration of suturing procedure, number of suture packs used during the suturing, subjective grading of suturing difficulty and need for extended suturing in operative room) | During suturing (from the delivery to one hour after the delivery)
  The duration of suturing procedure, number of suture packs used during the suturing, subjective grading of suturing difficulty and need for extended suturing in operative room
Postpartum symptoms two days after the delivery (Perineal pain evaluation using 11 points (0-10) Verbal Numeric Scale, urinary retention, perineal infection, perineal hematoma requiring surgical drainage, symptoms of urinary/anal incontinence) | During the second day after the delivery
  Perineal pain evaluation using 11 points (0-10) Verbal Numeric Scale, urinary retention (for more than 6 hours after the delivery/urinary catheter extraction), perineal infection, perineal hematoma requiring surgical drainage, symptoms of urinary/anal incontinence
Phone-call evaluation two months after the delivery | Two months after the delivery
  "Yes or no" questions regarding symptoms of urinary/anal incontinence, perineal complications (infection or dehiscence of perineal scar); timing of resumption of sexual activity; perineal pain and dyspareunia evaluation using 11 points (0-10) Verbal Numeric Scale.
Phone-call evaluation one year after the delivery (Two questionnaires) | One year after the delivery
  Two questionnaires will be filled: Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) and Pelvic Floor Distress Inventory-20 (PFDI-20)

CONTACTS AND LOCATIONS:
Overall Officials: Shlomi Sagi, M.D., Principal Investigator — Bnai-Zion Medical Center, Haifa, Israel; Reuven Keidar, M.D., Principal Investigator — Carmel Medical Center, Haifa, Israel; Ido Solt, M.D., Principal Investigator — Rambam Health Care Campus, Haifa, Israel; Asnat Walfisch, M.D., Principal Investigator — Hillel Yaffe Medical Center, Hadera, Israel; Dmitry Chuyun, M.D., Principal Investigator — The Baruch Padeh Medical Center, Poriya, Israel; David Peleg, M.D., Principal Investigator — Ziv Medical Center, Tzfat, Israel; Oleg Shnaider, M.D., Principal Investigator — Western Galilee Medical Center, Nahariya, Israel
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroli G, Mignini L. Episiotomy for vaginal birth. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD000081. doi: 10.1002/14651858.CD000081.pub2. PMID 19160176
- [Background] Pergialiotis V, Vlachos D, Protopapas A, Pappa K, Vlachos G. Risk factors for severe perineal lacerations during childbirth. Int J Gynaecol Obstet. 2014 Apr;125(1):6-14. doi: 10.1016/j.ijgo.2013.09.034. Epub 2014 Jan 9. PMID 24529800
- [Derived] Sagi-Dain L, Kreinin-Bleicher I, Bahous R, Gur Arye N, Shema T, Eshel A, Caspin O, Gonen R, Sagi S. Is it time to abandon episiotomy use? A randomized controlled trial (EPITRIAL). Int Urogynecol J. 2020 Nov;31(11):2377-2385. doi: 10.1007/s00192-020-04332-2. Epub 2020 May 24. PMID 32448935